CLINICAL TRIAL: NCT03126630
Title: Phase 1 Safety Run-In and Phase 2 Randomized Clinical Trial of Anetumab Ravtansine and Pembrolizumab (MK-3475) Compared to Pembrolizumab Alone for Mesothelin-Positive Malignant Pleural Mesothelioma
Brief Title: Pembrolizumab With or Without Anetumab Ravtansine in Treating Patients With Mesothelin-Positive Pleural Mesothelioma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00633; NCI-2017-00633 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1721; 10107 (Other: Dana-Farber - Harvard Cancer Center LAO); 10107 (Other: CTEP); UM1CA186686 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Pleural Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — anetumab ravtansine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Upon radiologic documentation of disease progression, patients may cross over to Group II.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Pharmacological Study
- Group II (anetumab ravtansine, pembrolizumab) (Experimental): Patients receive anetumab ravtansine IV over 1 hour and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 12 months for anetumab ravtansine and up to 24 months for pembrolizumab in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anetumab Ravtansine; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Pharmacological Study

INTERVENTIONS:
Biological: Anetumab Ravtansine — Given IV
  Other Names: BAY 94-9343
  Arms: Group II (anetumab ravtansine, pembrolizumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and how well pembrolizumab with or without anetumab ravtansine works in treating patients with mesothelin-positive pleural mesothelioma. Anetumab ravtansine is a monoclonal antibody, called anetumab, linked to a chemotherapy drug, called ravtansine. Anetumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as mesothelin receptors, and delivers ravtansine to kill them. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab and anetumab ravtansine may work better in treating patients with mesothelin-positive pleural mesothelioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose of anetumab ravtansine that is safe in combination with pembrolizumab to be used in the randomized phase 2 study. (Phase I safety lead-in) II. Determine if the overall response rate of the combination of anetumab ravtansine and pembrolizumab is superior to pembrolizumab alone. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the progression free survival of anetumab ravtansine and pembrolizumab compared to pembrolizumab alone.

II. To evaluate the pharmacodynamic effects of anetumab ravtansine and pembrolizumab on soluble megakaryocyte potentiating factor (MPF).

III. To evaluate the pharmacokinetics of anetumab ravtansine and pembrolizumab. IV. To evaluate mononuclear phagocyte system (MPS) function, FcgammaRs, hormone and chemokine mediators as methods to evaluate factors affecting the pharmacokinetics and pharmacodynamics of these agents.

V. To determine the incidence of antibodies directed against anetumab ravtansine.

CORRELATIVE STUDY OBJECTIVES:

I. To determine whether elevations in Bim in tumor-reactive T cells (TTR) predict responses to treatment and whether its detection is dynamic with treatment.

II. To determine whether soluble PD-L1 predicts responses to treatment and whether its detection is dynamic with treatment.

III. To evaluate PD-L1 expression in archival tissue as a predictive marker of response to pembrolizumab-based therapy.

IV. To explore the symptomatic adverse events (AE) for tolerability of each treatment group using Patient Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE).

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Upon radiologic documentation of disease progression, patients may cross over to Group II.

GROUP II: Patients receive anetumab ravtansine IV over 1 hour and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 12 months for anetumab ravtansine and up to 24 months for pembrolizumab in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION
* Patients must have histologically or cytologically confirmed malignant pleural mesothelioma
* Patient is willing to submit a tissue sample to test for expression of mesothelin

  * Note: Tissue sample for mesothelin assay may have been collected prior to, during or after receipt of the frontline chemotherapy; patients will not be required to submit another tissue sample after receipt of the chemotherapy
* Patients must have received platinum based chemotherapy
* REGISTRATION
* For phase 2 only:
* Patient has measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for non-pleural disease or modified RECIST 1.1 (mRECIST) for pleural disease

  * Note: For pleural disease, this is defined as at least one lesion that can be accurately measured perpendicular to the chest wall or mediastinum that is >= 10 mm (>= 1 cm); for extra pleural disease, measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 10 mm (>= 1 cm) for non-nodal lesions and >= 15 mm (>= 1.5 cm) for nodal lesions with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam as per RECIST 1.1
* Tissue submitted for testing at pre-registration shows moderate or stronger mesothelin expression in >= 30% of the tumor cells
* For phase 1 and 2:
* Patients must have received platinum-based therapy with or without bevacizumab
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN AND partial thromboplastin time (PTT) or activated PTT (aPTT) =< 1.5 x ULN, unless patient is on stable dose of anti-coagulation therapy in which case patients will be allowed to participate if they have no signs of bleeding or clotting and the INR/PT and PTT/aPTT results are compatible with an acceptable risk-benefit ratio as per the investigator's discretion
* Negative serum pregnancy test for females of child bearing potential

  * Note: Females are considered to not be of child bearing potential if any of the following apply:
  * Postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age, a high follicle stimulating hormone [FSH] level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient);
  * Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening;
  * Has a congenital or acquired condition that prevents childbearing
* Patient agrees to use one of the following acceptable methods of contraception prior to study entry, during study participation, and for at least six months after receiving the last dose of study treatment:

  * Acceptable methods of contraception are:

    * Single method (1 of the following is acceptable):

      * Abstinence, if consistently employed as the patient's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and Institutional Review Boards (IRBs)
      * Intrauterine device (IUD)
      * Vasectomy of a female patient's male partner
      * Contraceptive rod implanted into the skin
    * Combination method (requires use of 2 of the following):

      * Diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide)
      * Cervical cap with spermicide (nulliparous women only)
      * Contraceptive sponge (nulliparous women only)
      * Male condom or female condom (cannot be used together)
      * Hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin-only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection
* Ability to understand and the willingness to sign a written informed consent document, unless patient is of impaired decision making capacity in which case patient may be eligible if they have a legal authorized representative or caretaker available

Exclusion Criteria:

* Patients who have received any monoclonal antibody therapy within 4 weeks prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1)

  * Note: Patients with =< grade 2 neuropathy or =< grade 2 alopecia are an exception to this criterion and may qualify for the study
  * Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients who are receiving any other investigational agents
* Patients with known brain metastases with progressive neurologic dysfunction, requirement of steroids and lack of improvement on head imaging obtained prior to consent to this clinical trial should be excluded because of their poor prognosis and because they would confound the evaluation of neurologic and other adverse events

  * Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either magnetic resonance imaging [MRI] or computed tomography [CT] scan, for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
  * Note: Patients with carcinomatosis meningitis should also be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to anetumab ravtansine or pembrolizumab
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4, including herbal preparation containing CYP3A4 inducers (e.g., St. John's Wort), grapefruit and grapefruit juice (CYP3A4 inhibitor), within 2 weeks before the start of study treatment
* Patients are prohibited from receiving the following therapies during the screening and treatment phases (including retreatment for post-complete response relapse) of this trial:

  * Antineoplastic systemic chemotherapy or biological therapy
  * Immunotherapy not specified in this protocol
  * Chemotherapy not specified in this protocol
  * Investigational agents other than anetumab ravtansine and pembrolizumab
  * Radiation therapy (Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be considered on an exceptional case by case basis after consultation with Cancer Therapy Evaluation Program (CTEP); the patient must have clear measurable disease outside the radiated field; administration of palliative radiation therapy will be considered clinical progression for the purposes of determining progression free survival [PFS])
  * Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Chalmette-Guerin (BCG), and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
  * Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of suspected immunologic etiology; the use of physiologic doses of corticosteroids may be approved after consultation with the study principal investigator (PI) and CTEP
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or breastfeeding.

  * Note: Pregnant women are excluded from this study because anetumab ravtansine and pembrolizumab are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with anetumab ravtansine and pembrolizumab, breastfeeding should be discontinued if the mother is treated with anetumab ravtansine or pembrolizumab
* Human immunodeficiency virus (HIV)-positive patients who do not meet all of the following and/or are on HIV medications considered to be strong inhibitors or inducers of CYP3A4:

  * Undetectable HIV viral load by standard clinical assay within 6 months of registration
  * Willing to adhere to antiretroviral therapy that has minimal overlapping toxicity or pharmacokinetic interactions with protocol therapy
  * No acquired immunodeficiency syndrome (AIDS)-defining events other within the past 12 months
  * Near normal life expectancy if not for the presence of the cancer
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection

  * Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Patients who are known to have a history of or a finding of corneal epitheliopathy at pre-study are excluded because anetumab ravtansine may worsen this condition and reduce vision
* Known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
* Receipt of transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF], or recombinant erythropoietin) within 4 weeks prior to study treatment
* Patient with active interstitial lung disease (ILD)/pneumonitis or a prior history of ILD/pneumonitis requiring treatment with steroids
* Patient has received prior treatment with PD-1, PD-L1 or PD-L2 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2026-09-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Mansfield, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (33):
- United States (32):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2 Group I (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Upon radiologic documentation of disease progression, patients may cross over to Group II.
  >
  >
  >
  >
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  >
  >
  >
  >
  > Pembrolizumab: Given IV
  >
  >
  >
  >
  >
  > Pharmacological Study: Correlative studies
- Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab): Patients receive anetumab ravtansine IV over 1 hour and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 12 months for anetumab ravtansine and up to 24 months for pembrolizumab in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > Anetumab Ravtansine: Given IV
  >
  >
  >
  >
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  >
  >
  >
  >
  > Pembrolizumab: Given IV
  >
  >
  >
  >
  >
  > Pharmacological Study: Correlative studies
- Phase 1 Cohort Dose Level 1: Anetumab Ravtansine Dose 6.5 mg/kg
Period: Overall Study
Arm/Group | Phase 2 Group I (Pembrolizumab) | Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab) | Phase 1 Cohort Dose Level 1
Started | 18 | 18 | 13
Completed | 18 | 17 | 13
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 Group I (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Upon radiologic documentation of disease progression, patients may cross over to Group II.>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pembrolizumab: Given IV>
  >>
  >
  >> Pharmacological Study: Correlative studies
- Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab): Patients receive anetumab ravtansine IV over 1 hour and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 12 months for anetumab ravtansine and up to 24 months for pembrolizumab in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> Anetumab Ravtansine: Given IV>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pembrolizumab: Given IV>
  >>
  >
  >> Pharmacological Study: Correlative studies
- Phase 1 Cohort DLT 1: Anetumab Ravtansine & MK-3475: Anetumab ravtansine: Day 1 of each cycle for up to 12 months> MK-3475 (pembrolizumab): Day 1 of each cycle for up to 24 months
- Total: Total of all reporting groups
Arm/Group | Phase 2 Group I (Pembrolizumab) | Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab) | Phase 1 Cohort DLT 1: Anetumab Ravtansine & MK-3475 | Total
Number analyzed (Participants) | 17 | 18 | 13 | 48
Age, Continuous [Median (Full Range); unit: years] | 70.0 [46.0 to 85.0] | 67.5 [23.0 to 88.0] | 72 [48 to 81] | 68.0 [23.0 to 88.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 16
  Male | 11 | 12 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 17 | 5 | 38
  Unknown or Not Reported | 1 | 0 | 7 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 16 | 11 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Histologic Grade [Count of Participants; unit: Participants]
  Borderline malignancy | 0 | 1 | 0 | 1
  Grade cannot be assessed | 10 | 8 | 7 | 25
  Poorly Differentiated | 1 | 1 | 1 | 3
  Well Differentiated | 1 | 0 | 0 | 1
  Missing | 5 | 8 | 5 | 18
Disease Stage [Count of Participants; unit: Participants] — IA: Stage grouping (T1, N0, M0) or (T2, N0, M0)> IB: Stage grouping (T3, N0, M0)> II: Stage grouping (T1 or T2, N1, M0)> IIIA: Stage grouping (T3, N1, M0)> IIIB: Stage grouping (T1-T3, N2, M0) or (T4, Any N, M0)> IV: Stage grouping (Any T, Any N, M1)
  Participants
    Stage IA | 2 | 0 | 0 | 2
    Stage IB | 3 | 0 | 0 | 3
    Stage II | 0 | 1 | 1 | 2
    Stage III | 1 | 2 | 0 | 3
    Stage IIIB | 0 | 5 | 1 | 6
    Stage IV | 8 | 8 | 6 | 22
    Missing | 3 | 2 | 5 | 10
Weight [Mean (Full Range); unit: kg] | 77.2 [48.8 to 100.2] | 80.1 [53.2 to 108.0] | 85.0 [51.8 to 173] | 80.4 [48.8 to 173]
Height [Mean (Full Range); unit: cm] | 168.4 [152.8 to 188.0] | 173.1 [152.0 to 188.0] | 167.3 [90.9 to 196] | 169.2 [90.9 to 196]
BSA [Mean (Full Range); unit: m^2] — Body Surface Area
  m^2 | 1.9 [1.4 to 2.3] | 1.9 [1.6 to 2.3] | 1.9 [1.5 to 2.6] | 1.9 [1.4 to 2.6]
ECOG Performance Score [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status.> ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction. > ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. > ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. > ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 3 | 5 | 2 | 10
    1 | 14 | 13 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Phase 2 Confirmed Tumor Response Rate (Phase II)
Description: Will be assessed using Response Evaluation Criteria in Solid Tumors version 1.1 criteria. The proportion of successes will be estimated in each group by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated in each arm. Comparison of confirmed response rates between the two treatment groups will be performed using a one-sided z-test with pooled variance at significance level 0.10. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Group I (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Upon radiologic documentation of disease progression, patients may cross over to Group II.>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pembrolizumab: Given IV>
  >>
  >
  >> Pharmacological Study: Correlative studies
- Group II (Anetumab Ravtansine, Pembrolizumab): Patients receive anetumab ravtansine IV over 1 hour and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 12 months for anetumab ravtansine and up to 24 months for pembrolizumab in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> Anetumab Ravtansine: Given IV>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pembrolizumab: Given IV>
  >>
  >
  >> Pharmacological Study: Correlative studies
Arm/Group | Group I (Pembrolizumab) | Group II (Anetumab Ravtansine, Pembrolizumab)
Number analyzed (Participants) | 17 | 18
Participants
  NE | 2 | 4
  PD (Preliminary) | 6 | 2
  PD (Confirmed) | 3 | 1
  SD | 5 | 9
  PR (Confirmed) | 1 | 2
Statistical Analysis 1: Comparison: Group I (Pembrolizumab) vs Group II (Anetumab Ravtansine, Pembrolizumab); Test type: Equivalence — The null hypothesis that there are no differences between the classes in the population. The purpose of the test is to evaluate how likely the observed frequencies would be assuming the null hypothesis is true; p = 0.27541, Chi-squared

2. Primary Outcome: Phase I - Recommended Phase 2 Dose of Ametumab Ravtansine With Combination of Pembrolizumab
Description: All patients that have received any amount of the combination anetumab ravtansine and pembrolizumab will be evaluable for toxicity. Please note this is different from the definition of evaluable for dose-limiting toxicity (DLT) where patients who cannot complete the planned dose due to reasons other than toxicity will be replaced.
Time Frame: Up to 2 years
Measure: Number; unit: mg/kg IV
Groups:
- Phase 1 Cohort: Anetumab Ravtansine & MK-3475: Phase 1 Cohort: Anetumab ravtansine & MK-3475
Arm/Group | Phase 1 Cohort: Anetumab Ravtansine & MK-3475
Number analyzed (Participants) | 13
mg/kg IV | 6.5

3. Secondary Outcome: Phase 2 Duration of Response
Description: Will be defined as evaluable patients who achieved noted to be a partial response or complete response based Response Evaluation Criteria in Solid Tumors version 1.1 criteria. Will be estimated using the method of Kaplan-Meier. The comparison of duration of response between two treatment arms will be based on the log-rank test. This calculation will start with the date of start of treatment.
Time Frame: Up to 2 years
Population: Data were not collected and the outcome cannot be reported.
Groups:
- Group I (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Upon radiologic documentation of disease progression, patients may cross over to Group II.>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Pembrolizumab: Given IV>
  > Pharmacological Study: Correlative studies
- Group II (Anetumab Ravtansine, Pembrolizumab): Patients receive anetumab ravtansine IV over 1 hour and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 12 months for anetumab ravtansine and up to 24 months for pembrolizumab in the absence of disease progression or unacceptable toxicity.> > Anetumab Ravtansine: Given IV>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Pembrolizumab: Given IV>
  > Pharmacological Study: Correlative studies
Arm/Group | Group I (Pembrolizumab) | Group II (Anetumab Ravtansine, Pembrolizumab)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 2 Overall Survival
Description: Will be estimated using the method of Kaplan-Meier. The comparison of overall survival in event of death between two treatment arms will be based on the log-rank test.
Time Frame: From the start of treatment to death due to any cause, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pembrolizumab) | Group II (Anetumab Ravtansine, Pembrolizumab)
Number analyzed (Participants) | 17 | 18
Participants | 0 | 2
Statistical Analysis 1: Comparison: Group I (Pembrolizumab); Test type: Superiority; p = 0.1936, Log Rank; Hazard Ratio (HR) = 0.0, 95% CI 2-sided [lower limit 0.0] (Not enough events)

5. Secondary Outcome: Phase 2 Progression Free Survival
Description: Will be estimated using the method of Kaplan-Meier. The comparison of progression-free survival between two treatment arms will be based on the log-rank test. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the start of treatment to the earliest date of documentation of disease progression or death due to any cause, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pembrolizumab) | Group II (Anetumab Ravtansine, Pembrolizumab)
Number analyzed (Participants) | 17 | 18
Participants | 10 | 9
Statistical Analysis 1: Comparison: Group I (Pembrolizumab) vs Group II (Anetumab Ravtansine, Pembrolizumab); Test type: Superiority; p = 0.1952, Log Rank; Hazard Ratio (HR) = 1.81, 95% CI 2-sided [0.73 to 4.51]

6. Secondary Outcome: Pharmacokinetics of Anetumab Ravtansine
Description: Will be largely descriptive. Changes over time will be plotted and assessed for each patient.
Time Frame: Days 1 and 3 of courses 1 and 8
Reporting Status: Not Posted

7. Secondary Outcome: Change in Megakaryocyte Potentiating Factor Levels Assessed in Tumor
Description: Relative changes in biomarker levels will be compared by best overall response groups using the non-parametric Wilcoxon rank-sum test. Also, the associations between changes in megakaryocyte potentiating factor levels and ordered response categories (i.e. complete response-partial response-stable disease-progressive disease) will be assessed with the Jonckheere-Terpstra test for trend.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Mononuclear Phagocyte System -FcgammaRs and Chemokine Mediators of Mononuclear Phagocyte System
Description: The mean equivalent soluble fluorophore and antibody bound to cell (ABC) will be determined for each specimen. Linear regression will be used to explore the linear relationship between the continuous values of these mononuclear phagocyte system-FcgammaRs probes and anetumab ravtansine levels. The concentrations of CCL2 and CCL5 will be determined for each specimen. Linear regression will be used to explore the linear relationship between the continuous values of these chemokines and anetumab ravtansine levels.
Time Frame: Up to 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Incidence of Adverse Events
Description: To explore the symptomatic adverse events (AE) for tolerability of each treatment group using Patient Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Groups:
- Phase 2 Group I (Pembrolizumab); Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab): Pharmacological Study: Correlative studies
- Phase 1 Cohort DLT 1: Anetumab Ravtansine Dose 6.5 mg/kg
Arm/Group | Phase 2 Group I (Pembrolizumab) | Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab) | Phase 1 Cohort DLT 1
All-Cause Mortality (participants affected / at risk) | 1/17 | 2/18 | 1/13
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/18 | 1/13
Other Adverse Events (participants affected / at risk) | 17/17 | 18/18 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 Group I (Pembrolizumab) (N=17) | Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab) (N=18) | Phase 1 Cohort DLT 1 (N=13)
Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 Group I (Pembrolizumab) (N=17) | Phase 2 Group II (Anetumab Ravtansine, Pembrolizumab) (N=18) | Phase 1 Cohort DLT 1 (N=13)
Anemia (Blood and lymphatic system disorders) | 7 (42) | 7 (32) | 7 (54)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (9) | 4 (24) | 1 (12)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 6 (17) | 1 (2)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 2 (10) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (2) | 1 (1) | 2 (6)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (11) | 3 (14) | 3 (32)
Blurred vision (Eye disorders) | 0 (0) | 1 (8) | 2 (3)
Cataract (Eye disorders) | 0 (0) | 2 (12) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 0 (0) | 1 (9)
Dry eye (Eye disorders) | 2 (5) | 4 (28) | 2 (18)
Eye disorders - Other, specify (Eye disorders) | 2 (4) | 6 (73) | 3 (20)
Eye pain (Eye disorders) | 1 (3) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 2 (11) | 3 (20)
Uveitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 3 (11) | 4 (9)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (6) | 5 (12) | 6 (17)
Diarrhea (Gastrointestinal disorders) | 4 (8) | 11 (38) | 7 (26)
Dry mouth (Gastrointestinal disorders) | 1 (3) | 2 (8) | 3 (32)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (6) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (7) | 2 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (11)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (9) | 3 (16)
Nausea (Gastrointestinal disorders) | 3 (18) | 13 (62) | 6 (19)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 4 (7) | 3 (5)
Chills (General disorders) | 0 (0) | 2 (3) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 5 (19) | 2 (5)
Fatigue (General disorders) | 8 (58) | 12 (81) | 9 (48)
Fever (General disorders) | 2 (2) | 3 (7) | 2 (12)
Flu like symptoms (General disorders) | 0 (0) | 2 (3) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (2) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (3) | 0 (0) | 1 (2)
Malaise (General disorders) | 1 (6) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (4) | 3 (23) | 0 (0)
Pain (General disorders) | 4 (7) | 3 (10) | 2 (6)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (9) | 1 (4)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (3) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (8)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 2 (4) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Activated partial throm time prolonged (Investigations) | 1 (3) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 7 (35) | 7 (26)
Alkaline phosphatase increased (Investigations) | 4 (14) | 9 (22) | 7 (36)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 11 (65) | 8 (32)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 5 (19) | 4 (6) | 2 (10)
ECG QT corrected interval prolonged (Investigations) | 1 (14) | 3 (5) | 1 (3)
Investigations - Other, specify (Investigations) | 4 (14) | 7 (39) | 5 (42)
Lymphocyte count decreased (Investigations) | 6 (32) | 4 (18) | 6 (79)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (10) | 2 (3)
Platelet count decreased (Investigations) | 3 (4) | 4 (23) | 0 (0)
Weight loss (Investigations) | 3 (6) | 5 (17) | 1 (2)
White blood cell decreased (Investigations) | 1 (1) | 3 (10) | 2 (11)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (7) | 5 (21) | 7 (17)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 2 (5) | 2 (3)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (46) | 2 (5) | 4 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (7) | 1 (2) | 2 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (23) | 9 (32) | 5 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (11)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6) | 8 (21) | 3 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 4 (4) | 3 (3)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 5 (26) | 5 (23)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7) | 2 (10) | 4 (22)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (15) | 1 (20) | 3 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (14) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (14) | 0 (0) | 1 (2)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (3) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (15) | 5 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6) | 1 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (18) | 2 (7)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (6) | 4 (15) | 3 (9)
Hypersomnia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 0 (0) | 4 (15)
Paresthesia (Nervous system disorders) | 2 (16) | 2 (21) | 1 (9)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (14) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 9 (72) | 4 (48)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (14) | 3 (17) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 2 (18) | 1 (2)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (17) | 2 (7) | 6 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (41) | 7 (17) | 6 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (15)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (6) | 1 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (4) | 2 (12)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (12) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 1 (3)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 2 (9)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (14) | 0 (0) | 2 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 4 (11) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4) | 4 (17) | 2 (4)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (5) | 2 (3) | 3 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (9) | 3 (18)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3) | 1 (11)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (25) | 2 (2)
Hypotension (Vascular disorders) | 3 (7) | 1 (2) | 1 (4)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03126630/Prot_SAP_000.pdf